CLINICAL TRIAL: NCT06965413
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Trial to Assess Efficacy, Safety, and Tolerability of RO7204239 in Combination With Tirzepatide in Participants With Obesity or Overweight With At Least One Weight-related Comorbidity
Brief Title: A Study to Assess Efficacy, Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of RO7204239 in Combination With Tirzepatide in Participants With Obesity or Overweight With At Least One Weight-related Comorbidity
Acronym: GYMINDA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC45538; 2024-519561-22-00 (Registry Identifier: EU Trial Number)
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Overweight With One Weight Related Comorbidity
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo + Tirzepatide (Active Comparator): Participants will receive RO7204239 matching placebo via subcutaneous (SC) injection every 4 weeks (Q4W) for the core treatment period of 48 weeks and the treatment extension period of 24 weeks. Participants will also receive tirzepatide, as a background therapy, up-titrated according to the approved tirzepatide prescribing information, SC, every week (QW) during the core treatment period of 48 weeks.
  Interventions: Drug: RO7204239; Drug: RO7204239 Matching Placebo; Drug: Tirzepatide
- RO7204239 low dose + Tirzepatide (Experimental): Participants will receive RO7204239, low dose, SC, Q4W for the core treatment period of 48 weeks. During the treatment extension period participants will receive placebo for the period of 24 weeks. Participants will also receive tirzepatide, as a background therapy, up-titrated according to the approved tirzepatide prescribing information, SC, QW during the core treatment period of 48 weeks.
  Interventions: Drug: RO7204239; Drug: Tirzepatide
- RO7204239 medium dose + Tirzepatide (Experimental): Participants will receive RO7204239, medium dose, SC, Q4W for the core treatment period of 48 weeks. During the treatment extension period participants will receive placebo for the period of 24 weeks. Participants will also receive tirzepatide, as a background therapy, up-titrated according to the approved tirzepatide prescribing information, SC, QW during the core treatment period of 48 weeks.
  Interventions: Drug: RO7204239; Drug: Tirzepatide
- RO7204239 high dose + Tirzepatide (Experimental): Participants will receive RO7204239, high dose, SC, Q4W along with tirzepatide, given as a background therapy, up-titrated according to the approved tirzepatide prescribing information, SC, QW during the core treatment period of 48 weeks. During the treatment extension period participants will be randomized to receive RO7204239 or matching placebo, SC, Q4W for 24 weeks.
  Interventions: Drug: RO7204239; Drug: Tirzepatide

INTERVENTIONS:
Drug: RO7204239 — RO7204239 or matching placebo will be administered as per the schedule specified in the arms.
Drug: RO7204239 Matching Placebo — RO7204239 matching placebo will be administered as per the schedule specified in the arm.
  Arms: Placebo + Tirzepatide
Drug: Tirzepatide — Tirzepatide will be administered as per the schedule specified in the arms.

SUMMARY:
The main aim of the study is to assess the effect of RO7204239 in combination with tirzepatide, compared to placebo in combination with tirzepatide, on body weight loss after 48 weeks of treatment in adults with obesity or overweight with at least one weight-related comorbidity, but without diabetes mellitus (DM). The study comprises of a 4-week screening period; a 48-week core treatment period, where all participants will receive tirzepatide as background treatment and will be randomized to one of the 4 treatment arms; a 24-week treatment extension period, where participants will stop treatment with tirzepatide and a 24-week post-treatment follow-up (FU) period.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.0 kilograms per square meter (kg/m²) (additional weight-related comorbidities are not required for inclusion)
* BMI ≥ 27.0 kg/m² and < 30.0 kg/m² with at least one weight-related comorbidity such as: hypertension, dyslipidemia, obstructive sleep apnea and any cardiovascular disease
* History of at least one self-reported unsuccessful dietary or exercise effort to lose body weight
* Weight stability: self-reported change in body weight less than 5 kilograms (kg) (11 pounds [lbs]) within 3 months prior to screening

Exclusion Criteria:

* Prior history or diagnosis of DM
* Presence of non-proliferative diabetic retinopathy requiring acute therapy, proliferative diabetic retinopathy or diabetic macular edema
* Have obesity induced by other endocrinologic disorders
* Participation in unbalanced/extreme diets
* Prior or planned surgical treatment for obesity
* Endoscopic and/or device-based therapy for obesity or device removal within 6 months prior to screening
* Have a known clinically significant gastric emptying abnormality
* Have any of the following cardiovascular conditions within 6 months prior to screening: acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or hospitalization due to congestive heart failure (CHF)
* Have evidence of significant active, uncontrolled cardiovascular, autoimmune, endocrine, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, a neurological or psychiatric condition, or a history of any neuromuscular disorder or autoimmune/inflammatory disorders that may cause muscle wasting or medical condition capable of constituting a risk when taking the study medication or interfering with the interpretation of data, as judged by the investigator at screening
* Have evidence of a significant, uncontrolled endocrine abnormality
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy
* Have evidence of a significant, active autoimmune abnormality
* Have anemia
* Have signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2027-07-23 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight | Baseline, Week 48

SECONDARY OUTCOMES:
Absolute Change From Baseline in Body Weight | Baseline, Week 48
Change From Baseline in Body Mass Index (BMI) | Baseline, Week 48
Change From Baseline in Waist-to-height Ratio | Baseline, Week 48
Change From Baseline in Waist Circumference | Baseline, Week 48
Change From Baseline in Total Body Fat Mass Measured by Dual-energy X-ray Absorptiometry (DXA) | Baseline, Week 48
Change From Baseline in Total Lean Body Mass Measured by DXA | Baseline, Week 48
Change From Baseline in Appendicular Lean Mass Measured by DXA at Week 48 | Baseline, Week 48
Change From Baseline in Muscle Volume Measured by Magnetic Resonance Imaging (MRI) | Baseline, Week 48
Change From Baseline in Muscle Fat Infiltration Measured by MRI | Baseline, Week 48
Change From Baseline in Glycated Hemoglobin (HbA1C) Levels | Baseline, Week 48
Change From Baseline in Fasting Plasma Glucose Levels | Baseline, Week 48
Change From Baseline in Fasting C-peptide and Fasting Insulin Levels | Baseline, Week 48
Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, Week 48
Change From Baseline in Quantitative Insulin Sensitivity Check Index (QUICKI) | Baseline, Week 48
Change From Baseline in Fasting Lipid Profile | Baseline, Week 48
  Fasting lipid profile includes total cholesterol, triglycerides, low-density lipoprotein (LDL), high-density lipoprotein (HDL), non-HDL cholesterol
Number of Participants With Adverse Events (AEs) | Up to approximately 100 weeks
Number of Participants With Local and Systemic Injection Reactions | Up to approximately 100 weeks
Serum Concentrations of RO7204239 | Up to approximately 96 weeks
Steady-state Trough Concentration (Ctrough,ss) of RO7204239 | Up to approximately 96 weeks
Half-life (t1/2) of RO7204239 | Up to approximately 96 weeks
Steady-state Area Under the Concentration-time Curve Over One Dosing Interval (AUCtau,ss) of RO7204239 | Up to approximately 96 weeks
Steady-state Maximum Concentration (Cmax,ss) of RO7204239 | Up to approximately 96 weeks
Apparent Clearance (CL/F) of RO7204239 | Up to approximately 96 weeks
Apparent Volume of Distribution (Vd/F) of RO7204239 | Up to approximately 96 weeks
Number of Participants With Anti-drug Antibodies (ADAs) to RO7204239 | Up to approximately 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (19):
  - Pinnacle Research Group, Anniston, Alabama
  - Encompass Clinical Research, Spring Valley, California
  - K2 Medical Research-Winter Garden, Clermont, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Accellacare of Duly Health and Care, Oak Lawn, Illinois
  - Rochester Clinical Research, Rochester, New York
  - Accellacare of Salisbury, Salisbury, North Carolina
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - Accellacare of Wilmington, LLC, Wilmington, North Carolina
  - Accellacare Research of Winston Salem, Winston-Salem, North Carolina
  - NexGen Research, Lima, Ohio
  - Accellacare of Bristol/ Internal Medicine & Pediatrics, Bristol, Tennessee
  - Accellacare of Knoxville, Knoxville, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Juno Research, LLC, Houston, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Velocity Clinical Research (Impact Research Institute), Waco, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
- Poland (4):
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne ALL-MED, Krakow
  - Ekamed sp. z o.o., Lublin
  - ETG Warszawa, Warsaw
- Spain (6):
  - Universidad de Sevilla - Hospital Universitario Virgen Macarena, Seville, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Vithas Nisa Sevilla, Castilleja de la Cuesta, Granada
  - Hospital San Rafael A Coruna, A Coruña, LA Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
- United Kingdom (6):
  - Fylde Coast Clinical Research at Layton Medical Centre, Blackpool, Lancashire
  - University Hospitals of Leicester NHS Trust - Leicester General Hospital (LGH), Leicester, Leicestershire
  - Accellacare Yorkshire, Shipley, Yorkshire
  - Accellacare Warwickshire, Coventry
  - Accellacare North London, Northwood
  - Accellacare South London, Orpington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing